CLINICAL TRIAL: NCT00743886
Title: Influence of PRGF on Healing of MCL Tear - Randomized-Double-Blind-Placebo Control Trail
Brief Title: Influence of Plasma Rich in Growth Factors (PRGF) on Healing of Medial Collateral Ligament (MCL) Tear
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Omer Mei-Dan, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5000
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: MCL Tear
MeSH Terms: interventions — Intercellular Signaling Peptides and Proteins; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): saline
  Interventions: Drug: saline
- 1 (Experimental): Plasma Rich in Growth Factors (PRGF)
  Interventions: Biological: Plasma Rich in Growth Factors (PRGF)

INTERVENTIONS:
Biological: Plasma Rich in Growth Factors (PRGF) — injection onto injured area in ligament dose: 3-6mg
  Other Names: platelet-derived preparation rich in growth factors
  Arms: 1
Drug: saline — injection of 6 cc of saline into injured area
  Other Names: saline 0.9% NaCl
  Arms: 2

SUMMARY:
To evaluate the influence of Plasma Rich in Growth Factors (PRGF) on the healing process of medial collateral ligament (MCL) tear.

DETAILED DESCRIPTION:
Autologous platelet-rich matrices may aid in the healing of ligaments & tendons by promoting and accelerating tissue healing because of the release of growth factors including transforming growth factor (TGF)-beta1 and platelet-derived growth factor (PDGF) from platelet alpha-granules.

ELIGIBILITY:
Inclusion Criteria:

* age 18-40 years old
* diagnosed MCL tear grade 2/3

Exclusion Criteria:

* pregnancy
* mental or physical disabilities

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
time and efficiency of healing | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Omer Mei Dan, Dr, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel